CLINICAL TRIAL: NCT06382675
Title: Clinical Performance of the New Plasma Filter PX2 in Combination with the MultiFiltrate and MultiFiltratePRO in TPE Treatments
Brief Title: Clinical Performance of the New Plasma Filter PX2 in TPE Treatments
Acronym: plasmaFlux
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: KLIFO GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-PF-01-DE; CIV-23-11-044643 (Other: Unique identification number EUDAMED)
Record Dates: First submitted 2024-02-22; First posted 2024-04-24 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Autoimmune Diseases
Keywords: Therapeutical Plasma Exchange
MeSH Terms: conditions — Autoimmune Diseases | interventions — Plasma Exchange

STUDY DESIGN:
Intervention Model Description: Interventional, single arm, multi-centric, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapeutic Plasma Exchange (TPE) (Other): Patients with indication for TPE treatment according to American Society for Apheresis (ASFA) guideline
  Interventions: Device: Therapeutic Plasma Exchange (TPE) with the Plasma Filter PX2

INTERVENTIONS:
Device: Therapeutic Plasma Exchange (TPE) with the Plasma Filter PX2 — 230 evaluable TPE treatments will be documented in the study (with an average of 5-7 TPE treatments per patient this corresponds to approximately 46 patients)

SUMMARY:
The plasma filter is applied for a single use in extracorporeal blood purification therapy. The intended purpose is the separation of plasma from blood by filtration, in conditions, which are associated with increased concentration of plasma components where a rapid depletion slows down or stops a pathogenic process.

The investigation involves the collection of treatment data of the new Plasma Filter PX2 in combination with the multiFiltrate and multiFiltratePRO in therapeutic plasma exchange (TPE) treatments. The multiFiltrate and multiFiltratePRO are devices for extracorporeal blood purification treatments. No further control treatments will be investigated in this one arm design. The design is considered to be appropriate to reflect daily clinical practice and to contribute to empirical evidence of performance of the new Plasma Filter PX2. No specific treatment schedule is defined by the study protocol. The TPE treatment is performed with the plasma filter PX2 (investigational device) according to clinical practice established in each of the participating centers and are prescribed at the discretion of the treating physician. The participation in the study will have no influence on the treatment plan. The documentation of the treatment includes the therapy up to the tenth (10th) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by study patient and investigator/authorized physician
* Minimum age of 18 years
* Patients with an indication for a therapeutical plasma exchange
* Patients to be treated with the plasma filter PX2 in combination with the multiFiltrate or multiFiltratePRO
* No contraindication against systemic anticoagulation
* Ability to understand the nature and requirements of the study

Exclusion Criteria:

* Patients with known or suspected hypersensitivity to any of the materials of the PX2 plasma filter (Polysulfone, Polyvinylpyrrolidone, Polypropylene, Polyurethane, Silicone) and trial related products
* Patients suffering from a heparin allergy
* Patients with a prescription for TPE treatment with the completion of < 0.8 PV and > 2.0 PV
* Any conditions which could interfere with the patient's ability to comply with the study
* Women of childbearing age (< 55 years) without effective means of contraception, pregnancy (pregnancy test will be conducted at start) or lactation period
* Participation in a different interventional clinical study during the preceding 30 days
* Previous participation in this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Analysis of TPE treatments with the Plama Filter PX2 | on average 7 weeks depending on on the indication, frequency and number of treatments
  Investigation of clinical performance of the new plasma filter PX2 by assessing the completion of the prescribed plasma volume (PV) in ≥ 75% of all TPE procedures

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Büttner, Dr. med., Principal Investigator — Klinikum Aschaffenburg-Alzenau
Locations (5):
- Germany (5):
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg, Bavaria
  - Klinikum der Ludwig-Maximilians-Universität München (LMU Klinikum), Munich, Bavaria
  - Städtisches Klinikum Braunschweig, Braunschweig, Lower Saxony
  - St. Vincenz Kliniken, Paderborn, North Rhine-Westphalia
  - Charité-Universitätsmedizin Berlin, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: No